CLINICAL TRIAL: NCT02731001
Title: Proton Therapy to Reduce Acute Normal Tissue Toxicity in Locally Advanced Non-small-cell Lung Cancer
Acronym: PRONTOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other); National Center for Radiation Research in Oncology Dresden/Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Esther Troost, Prof. Esther Troost, Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR - PRONTOX - 2014
Record Dates: First submitted 2016-04-01; First posted 2016-04-07 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proton therapy (Experimental): Patients within the proton arm will receive 66 Gy(RBE) delivered with 6 fractions per week.
  Interventions: Radiation: Proton therapy
- Photon therapy (Active Comparator): Patients within the photon arm will be treated by intensity modulated radiotherapy with 6 fractions per week to a total dose of 66 Gy.
  Interventions: Radiation: Photon therapy

INTERVENTIONS:
Radiation: Proton therapy
  Arms: Proton therapy
Radiation: Photon therapy
  Arms: Photon therapy

SUMMARY:
The aims of the study are to reduce acute radiation induced side effects, i.e. pneumonitis and esophagitis grade II or higher by the use of proton therapy compared to photon radiotherapy of equal total dose. Secondary endpoints include evaluation of quality of life, loco-regional control, survival and late radiation induced side effects.

DETAILED DESCRIPTION:
Patients in this trial undergo primary radiochemotherapy for locally advanced NSCLC. As early and intermediate late effects of radiotherapy do not only hamper quality of life but can, in the case of radiation induced pneumonitis, be potentially lethal, a reduction of these side effects is desirable. Patients in this trial are 1:1 randomised to intensity modulated radiotherapy with photons or proton therapy. The primary aim of the study is to show a decrease of pneumonitis and or esophagitis grade 2 or higher by proton therapy. The observed incidence of both these side effects is 39% with photon therapy. The estimated incidence with proton therapy is around 12 %. Simultaneous chemotherapy will be applied to current clinical standards.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC (confirmed by cytology or histology) staged UICC IIIA or IIIB or UICC II if the patient declines surgery
* no distant metastases (M1)
* patient' age between 18 and 70 years
* Patient medically suited for primary radiochemotherapy with curative intent
* signed declaration of informed consent
* adequate compliance for treatment and clinical follow up
* adequate contraception during and after therapy if indicated

Exclusion Criteria:

* Participation in other interventional trial
* T1 or T2 N0 tumours that are candidates for stereotactic radiotherapy
* relevant neurological or psychiatric disorders that hinder treatment, follow-up or understanding of the procedures
* pregnant or breastfeeding women
* prior thoracic radiotherapy
* history of other malignancies during the last 5 years (exceptions can be made for tumours with excellent outcome)
* weight loss greater than 15% before therapy
* serological alterations (liver, kidney) prohibiting application of simultaneous chemotherapy
* respiratory motion of the tumour > 10 mm (evaluated by 4D CT), also when methods for motion reduction (abdominal compression) are used

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2016-08; Primary Completion 2021-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of acute and intermediate radiation induced side effects | no later than six months after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Esther Troost, Prof., Study Chair — Technische Universität Dresden, German Cancer Consortium, Helmholtz-Zentrum Dresden - Rossendorf
Locations (1):
- Department of Radiotherapy and Radiation Oncology, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zschaeck S, Simon M, Lock S, Troost EG, Stutzer K, Wohlfahrt P, Appold S, Makocki S, Butof R, Richter C, Baumann M, Krause M. PRONTOX - proton therapy to reduce acute normal tissue toxicity in locally advanced non-small-cell lung carcinomas (NSCLC): study protocol for a randomised controlled trial. Trials. 2016 Nov 15;17(1):543. doi: 10.1186/s13063-016-1679-4. PMID 27846903